CLINICAL TRIAL: NCT06312592
Title: Owning Rights and Protection: GBV Prevention, Mitigation, and Response in Colombia
Brief Title: GBV Prevention, Mitigation, and Response in Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Universidad de Los Andes (Unknown)
Responsible Party: Principal Investigator, Lindsay Stark, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWA00015367
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Refugee Self-reliance; Mental Health Issue; Empowerment; Gender Based Violence Knowledge and Perceived Risk; Decision Making
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receives the Entrepreneurship School with Gender Lens intervention. Participants receive a general training with six modules focused on business modeling and female empowerment for the participants. It is targeted for women who are forcibly displaced people, including refugees, and who are survivors or at risk of Sexual or Gender Based Violence. Each women entrepreneur, participates in individual mentoring sessions to build their business plan after the training and receives $800 start-up capital for their business plan. For at least a year, entrepreneurs will have a follow-up to promote their business scale up, including how to formalize their business in the market, how to define new strategies, and how to answer to the market's evolving requirements. Additionally, the participants receive an extensive training in gender aspects that have been identified as relevant to promote women's empowerment. The intervention also includes mental health content.
  Interventions: Behavioral: Entrepreneurship School with Gender Lens
- Control group (No Intervention): Does not receive the Entrepreneurship School with Gender Lens intervention the Entrepreneurship School with Gender Lens intervention

INTERVENTIONS:
Behavioral: Entrepreneurship School with Gender Lens — The Entrepreneurship School with Gender Lens (ESGL) is an approach that targets gender based violence survivors and women at-risk to help them develop business ideas, access needed support for the prevention of and response to GBV, exploitation and trafficking, and improve participants' overall self-reliance. Participants will go through a general business curriculum, work on business plans and learn gender issues and ways to mitigate GBV risks. Upon training completion, participants are eligible to pitch their business idea to a panel of experts and receive $800 of seed capital. They will also receive follow-up business advisory support for at least six months, focusing on access to markets and finance and building support networks, in order to continue building self-reliance.
  The ESGL will also include a mental health and psychosocial support module.
  Arms: Intervention group

SUMMARY:
As of August 2021, Colombia hosts the vast majority of Venezuelan refugees and migrants (UNHCR, 2022). For vulnerable refugees and migrants in Colombia, and especially for women, gender-based violence (GBV) is present during transit and continues in their new homes where xenophobia, lack of accessible and adequate services, lack of safe economic opportunities, and lack of information on access to services, further increase risk. Lack of livelihood opportunities also affect vulnerable refugees and migrants, especially women, with barriers to employment including lack of information; precarious working conditions with lower payments and longer working days with increasing risks of labor exploitation; xenophobia and discrimination; limited access to formal labor markets; lack of access to financial services, among others. To address these issues, the investigators are conducting a pilot randomized-controlled trial (RCT) of HIAS' Entrepreneurship School with Gender Lens (ESGL), a methodology that targets GBV survivors and women at-risk to help them develop business ideas, access needed support for the prevention of and response to GBV, exploitation and trafficking, and improve participants' overall self-reliance. The pilot RCT will be conducted within three cities in Colombia; approximately 80 eligible participants will be enrolled in each city and randomized to a treatment or control arm. Survey questionnaires will be administered to participants at baseline, eight months following baseline (endline), and 3-4 months after endline. Outcomes of interest include household self-reliance, mental health, empowerment, decision-making, and GBV risk and knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* At least 18 years of age
* At risk of gender based violence (GBV) or ever experienced GBV
* Have a migratory permit (for migrants/refugees)
* Colombian or Venezuelan, living in Colombia for at least six months
* Hold an entrepreneur profile registered with HIAS (the implementing partner).

Exclusion Criteria:

* Man or does not self identify as a woman
* Less than 18 years old
* Not at risk of GBV and never experienced GBV
* Does not have a migratory permit
* Not Colombian or Venezuelan
* Living in Colombia for less than six months
* No entrepreneur profile registered with HIAS (the implementing partner).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self identification
Enrollment: 253 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Los Andes University, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified by HIAS through existing databases, external referrals from other organizations in the field and open calls. Potential participants were then prescreened, screened, and enrolled in the study based on a set of criteria from March 11th to 21st, 2024.
Pre-assignment Details: Of 286 individuals screened, 253 met inclusion criteria and were randomized to treatment.
Groups:
- Intervention Group: Entrepreneurship School with Gender Lens: The Entrepreneurship School with Gender Lens (ESGL) is an approach that targets gender based violence survivors and women at-risk to help them develop business ideas, access needed support for the prevention of and response to GBV, exploitation and trafficking, and improve participants' overall self-reliance. Participants will go through a general business curriculum, work on business plans and learn gender issues and ways to mitigate GBV risks. Upon training completion, participants are eligible to pitch their business idea to a panel of experts and receive $800 of seed capital. They will also receive follow-up business advisory support for at least six months, focusing on access to markets and finance and building support networks, in order to continue building self-reliance.
  The ESGL also includes a mental health and psychosocial support module.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 175 | 78
Completed | 146 | 65
Not Completed | 29 | 13
Not completed — Lost to Follow-up | 29 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 175 | 78 | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 169 | 76 | 245
  >=65 years | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.50 (11.49) | 39.04 (12.12) | 39.36 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 78 | 253
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 175 | 78 | 253
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 175 | 78 | 253
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Colombia | 175 | 78 | 253
Self-Reliance Index [Mean (Standard Deviation); unit: units on a scale] | 3.27 (0.56) | 3.27 (0.50) | 3.27 (0.54)
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] | 7.66 (5.25) | 9.01 (4.82) | 8.08 (5.15)
Brief Resilient Coping Scale [Mean (Standard Deviation); unit: units on a scale] | 16.85 (2.18) | 16.85 (1.41) | 16.85 (1.97)
Completed primary school [Count of Participants; unit: Participants] | 123 | 60 | 183
Household size [Mean (Standard Deviation); unit: people] | 4.05 (1.61) | 4.18 (1.79) | 4.09 (1.66)
Nationality [Count of Participants; unit: Participants] — Participant nationality. All participants are either Colombian or Venezuelan.
  Participants
    Colombian | 51 | 21 | 72
    Venezuelan | 124 | 57 | 181

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reliance Index From Baseline to Endline
Description: The Self-Reliance Index (SRI) is a measure of refugee self-reliance, created by the Refugee Self-Reliance Initiative. The final score is calculated using 12 domains of self-reliance, including the health-related domains of healthcare access and health status. SRI scores may assume a value from 1 to 5, with 5 indicating greater self-reliance.
Time Frame: Past three months
Population: The sample that was measured at both baseline and endline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 146 | 65
score on a scale | -0.03 (0.64) | -0.21 (0.66)

2. Secondary Outcome: Change in Patient Health Questionnaire (PHQ-9) Score From Baseline to Endline
Description: The Patient Health Questionnaire (PHQ-9) is a 9-item measure of depression. The score may assume a value from 0 to 27, with higher scores signaling greater depressive symptomology.
Time Frame: Past two weeks
Population: Participants measured at baseline and endline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 146 | 65
score on a scale | -0.93 (5.21) | -1.49 (5.71)

3. Secondary Outcome: Change in Brief Scale of Resilient Strategies From Baseline to Endline
Description: The BriefScale of Resilient Strategies is a 4-item measure of resilience. The score may assume a value from 4 to 20, with higher scores signaling greater resilience.
Time Frame: Last three months
Population: Participants who were measured at baseline and endline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 146 | 65
score on a scale | 1.10 (3.35) | 0.43 (3.66)

ADVERSE EVENTS:
Time Frame: Eight months
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/78
Other Adverse Events (participants affected / at risk) | 0/175 | 0/78

LIMITATIONS AND CAVEATS:
The study was originally designed to include a third round of data collection for March 2025. However, the study received a stop work order and termination from the funder in January 2025, preventing the last round of data collection from taking place. As such, the study is a pilot RCT with baseline and endline data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT06312592/Prot_001.pdf
  • Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT06312592/SAP_002.pdf
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT06312592/ICF_000.pdf